CLINICAL TRIAL: NCT04744012
Title: Modified Periostal Pocket Flap Technique: a Case Series
Brief Title: Modified Periostal Pocket Flap Technique
Status: Completed | Type: Observational
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Jesús Torres García Denche, Associate Professor, Universidad Complutense de Madrid
Other Study IDs: P-15/568
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Bone Regeneration
Keywords: Periostal Pocket Flap Technique; PPFT

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- unique group: After local anesthesia, a full thickness flap was elevated from the lingual wall and a partial thickness flap was performed in the buccal one. After that, the buccal periosteum was detached and dental implants were placed following the biological drilling protocol, getting autologous bone particles from the implant site.
  Patient's blood collection was performed and the plasm obtained was poured down on a sterile container and mixed with autologous bone particles collected previously during the drilling procedure. Finally the graft was placed in the pocket prepared previously and the surgical wound was sutured in two planes.
  Interventions: Procedure: Modified Periostal Pocket Flap Technique

INTERVENTIONS:
Procedure: Modified Periostal Pocket Flap Technique — After local anesthesia, a full thickness flap was elevated from the lingual wall and a partial thickness flap was performed in the buccal one. After that, the buccal periosteum was detached and dental implants were placed following the biological drilling protocol, getting autologous bone particles from the implant site.
  Patient's blood collection was performed and the plasm obtained was poured down on a sterile container and mixed with autologous bone particles collected previously during the drilling procedure. Finally the graft was placed in the pocket prepared previously and the surgical wound was sutured in two planes.

SUMMARY:
The aim of this study is to propose a modification of the original periostal pocket flap technique consisting in replacing the xenograft by a conglomerate which contains autologous bone obtained from the future implant site through biological drilling technique and PRGF (Plasma Rich in Growth Factors)

DETAILED DESCRIPTION:
Materials and methods: 8 patients referred for implant placement and with a slight bucco-lingual (BL) width deficiency in alveolar bone were included in the study. Patients were placed dental implants and bone width was augmented by using the conglomerate mentioned above.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a favorable bone density and favorable bone length but insufficient bone width that could compromise implant placement

Exclusion Criteria:

* Smokers (>10 cigarettes per day) and patients with severe systemic disease ( ASA III or IV - American Society of Anaesthesiology)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients included in this case series were collected from Clinica Dental Alcalá, were operated on by the same surgeon and fullfilled the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2016-09-11 (Actual); Primary Completion 2016-09-24 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Volume of bone augmentation | 4 months
  Volume of bone augmentation of the surgical sites was measured in the postoperative parasagittal CT scans using a region of interest (ROI) containing the entire bone box regenerated area using the closed polygon tool of the OsiriX software

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Torres, Associate, Principal Investigator — Universidad Complutense de Madrid

IPD SHARING:
Plan to Share IPD: No